CLINICAL TRIAL: NCT02295995
Title: Exercise as an Adjuvant Therapy for Veterans With PTSD
Brief Title: Exercise and PTSD in Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D1316-W; 5IK2RX001316-02 (NIH); 1IK2RX001316-01A2 (NIH)
Record Dates: First submitted 2014-10-27; First posted 2014-11-20 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Post-traumatic
Keywords: Aged; Exercise; Veterans; Adherence; Clinical Trials, Randomized
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity (Experimental): Participants randomized to this arm will be enrolled in a 12-week physical activity program.
  Interventions: Behavioral: Exercise as an Adjuvant Therapy for Veterans with PTSD
- Usual Care Wait-List (No Intervention): Participants randomized to this arm will continue to receive usual care services for PTSD through the Veterans Health Administration (VHA) for 12 weeks after which time they will be offered the physical activity program for 12 weeks.

INTERVENTIONS:
Behavioral: Exercise as an Adjuvant Therapy for Veterans with PTSD — Methods: Approximately 50 Veterans 60 years and older with PTSD will be recruited to participate in a 12-week physical activity program consisting of aerobic and strength-training activities. Participants will be randomized to an intervention arm or usual care wait-list control. Outcomes: Changes in physical function, PTSD symptom severity, and aerobic endurance will be assessed between the two study arms. Secondary outcomes include compliance with the intervention, pain, sleep, and psychological well-being.
  Arms: Physical Activity

SUMMARY:
The purpose of this study is to examine whether posttraumatic stress disorder (PTSD) symptoms impact adherence to a 12-week physical activity program and whether exercise can help improve PTSD symptoms and health outcomes in older Veterans. Veterans over the age of 60 with PTSD were be recruited to participate in a 12-week physical activity program consisting of aerobic and strengthening activities. 54 participants were randomized to an intervention arm (n=36) or usual care wait-list control (n=18).

DETAILED DESCRIPTION:
There is substantial evidence that physical inactivity contributes to poorer physical health outcomes in older adults. There is a paucity of work examining physical activity in Veterans with PTSD. Consequently, the efficacy of exercise as a beneficial adjunctive therapy in the treatment for PTSD symptoms and related health sequelae has not been established. Methods: Approximately 50 Veterans 60 years and older with PTSD will be recruited to participate in a 12-week physical activity program consisting of aerobic and strength-training activities. Participants will be randomized to an intervention arm or usual care wait-list control. Outcomes: Changes in physical function, PTSD symptom severity, and aerobic endurance will be assessed between the two study arms. Summary: This pilot trial will extend the investigators' understanding of the physical and psychological benefits of physical activity in Veterans with PTSD. The results from this study will be used to be used to develop a larger, randomized controlled exercise trial for Veterans with PTSD. Once new, effective exercise therapies for Veterans with PTSD are established, we can augment traditional PTSD therapy with exercise therapy to promote the prevention and treatment of chronic diseases common in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for current PTSD,
* live within 50 miles of Durham VA Medical Center (VAMC) and have reliable transportation,
* registered for care at the Durham VAMC,
* independently mobile (assistive devices acceptable),
* speak and write fluent conversational English

Exclusion Criteria:

* Active substance dependence other than nicotine,
* cognitive impairment, uncontrolled psychotic symptoms,
* clinical history of cardiovascular disease (CVD) occurring within the past 3 months,
* uncontrolled hypertension,
* renal disease or currently receiving dialysis,
* psychotropic medication initiated within 6 weeks prior to enrollment
* proliferative retinopathy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Shepherd Hall, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall KS, Morey MC, Beckham JC, Bosworth HB, Pebole MM, Pieper CF, Sloane R. The Warrior Wellness Study: A Randomized Controlled Exercise Trial for Older Veterans with PTSD. Transl J Am Coll Sports Med. 2018 Mar 15;3(6):43-51. doi: 10.1249/TJX.0000000000000056. PMID 29632895
- [Result] Pebole MM, Hall KS. Physical activity promotion in women with PTSD: What we need for progress. Psychol Sport Exerc. 2019 Mar;41:127-129. PMID 31057332
- [Result] Hall KS, Morey MC, Bosworth HB, Beckham JC, Pebole MM, Sloane R, Pieper CF. Pilot randomized controlled trial of exercise training for older veterans with PTSD. J Behav Med. 2020 Aug;43(4):648-659. doi: 10.1007/s10865-019-00073-w. Epub 2019 Jul 1. PMID 31264055
- See also: Click here for more information about this study: Exercise as an Adjuvant Therapy for Veterans with PTSD — https://www.research.va.gov/currents/0418-Older-Veterans-with-PTSD-take-part-in-exercise-program.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: Participants randomized to this arm were enrolled in a 12-week, supervised exercise program.
- Usual Care Wait-List: Participants randomized to this arm continued to receive usual care services for PTSD through the Veterans Health Administration (VHA) for 12 weeks after which time they will be offered the physical activity program for 12 weeks.
Period: Overall Study
Arm/Group | Exercise | Usual Care Wait-List
Started | 36 | 18
Completed | 31 | 17
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Wait-List: Participants randomized to this arm continued to receive usual care services for PTSD through the VHA for 12 weeks after which time they will be offered the physical activity program for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Exercise | Usual Care Wait-List | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (3.2) | 66.9 (4.3) | 67.3 (3.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 34 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 18 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 13 | 46
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
PTSD Checklist DSM-V (PTSD symptoms) [Mean (Standard Deviation); unit: units on a scale] — This scale measures PTSD symptoms. Total scale range from 0 to 80, with higher scores indicating more severe PTSD symptoms
  units on a scale | 42.9 (14.9) | 41.1 (14.0) | 42.0 (14.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (5.9) | 30.4 (4.4) | 30.5 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Patient Recruitment
Description: The primary aim/outcome of this pilot study is the feasibility of recruiting older Veterans with PTSD to participate in a 12-week exercise program. The number of Veterans recruited out of the total number contacted will be determined at baseline.
Time Frame: Baseline
Population: 701 potentially eligible patients were identified, of which 380 were screened out. Leaving 321 eligible patients (the denominator). Of these 321, 168 declined participation, and 99 were unable to contact; leaving 54 that were enrolled/randomized (numerator).
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Number of potentially eligible patients contacted to participate in the study.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 321
Participants | 54

2. Primary Outcome: Physical Activity
Description: Activity levels (metabolic equivalent [MET]-minutes/week) were measured using the Aerobic Center Longitudinal Study physical activity questionnaire.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Error); unit: metabolic equivalent (MET)-min/week
Arm/Group | Exercise | Usual Care Wait-List
Number analyzed (Participants) | 31 | 17
metabolic equivalent (MET)-min/week
  Baseline | 365.8 (349.4) | 349.4 (122.2)
  12 Weeks | 1954.4 (192.2) | 675.3 (178.8)
Statistical Analysis 1: Comparison: Exercise vs Usual Care Wait-List; The between-group difference at 12 weeks [mean difference (MD) and 95% Confidence Interval] was calculated for all outcome measures. Cohen's d effect sizes were calculated as the difference in mean-level change (from baseline to 12 weeks) between the two groups divided by the standard deviation (SD) and is interpreted as d=0.20 (small), d=0.50 (medium), and d=0.80 (large). Cohen's d for physical activity in this sample was 1.37; Test type: Other; Cohen's d calculated as the change from baseline to 12 weeks in both groups

3. Primary Outcome: PTSD Symptoms
Description: PTSD symptom severity was assessed at both baseline and 12 Weeks using the PTSD Checklist for DSM-V (PCL-5). Scores on the PCL-5 range from 0 to 80, with higher scores indicating more severe PTSD symptoms.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Exercise | Usual Care Wait-List
Number analyzed (Participants) | 31 | 17
score on a scale
  Baseline | 42.97 (2.5) | 41.06 (3.5)
  12 Weeks | 35.87 (2.4) | 38.19 (2.3)
Statistical Analysis 1: Comparison: Exercise vs Usual Care Wait-List; The between-group difference at 12 weeks [mean difference (MD) and 95% Confidence Interval] was calculated for all outcome measures. Cohen's d effect sizes were calculated as the difference in mean-level change (from baseline to 12 weeks) between the two groups divided by the standard deviation (SD) and is interpreted as d=0.20 (small), d=0.50 (medium), and d=0.80 (large). Cohen's d for PCL-5 in this sample was 0.38; Test type: Other; Cohen's d calculated as the change from baseline to 12 weeks in both groups

4. Secondary Outcome: Aerobic Endurance
Description: Aerobic endurance was assessed using the 6-minute walk test (distance).
Time Frame: Baseline and 12 Weeks
Population: 2 participants in the usual care (UC) condition did not complete this test at 12 weeks, and were not included in this analysis.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Exercise | Usual Care Wait-List
Number analyzed (Participants) | 31 | 15
meters
  Baseline | 462.1 (22.3) | 465.9 (32.0)
  12 Weeks | 531.1 (29.8) | 476.0 (21.7)
Statistical Analysis 1: Comparison: Exercise vs Usual Care Wait-List; The between-group difference at 12 weeks [mean difference (MD) and 95% Confidence Interval] was calculated for all outcome measures. Cohen's d effect sizes were calculated as the difference in mean-level change (from baseline to 12 weeks) between the two groups divided by the standard deviation (SD) and is interpreted as d=0.20 (small), d=0.50 (medium), and d=0.80 (large). Cohen's d for 6-minute walk in this sample was 0.50; Test type: Other; Cohen's d calculated as the change from baseline to 12 weeks in both groups

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for 12 weeks (the duration of the intervention period).
Groups:
- Exercise: Participants randomized to this arm were enrolled in a 12-week, supervised exercise program. 36 patients were randomized, of which 31 completed the intervention (included in analyses).
- Usual Care Wait-List: Participants randomized to this arm continued to receive usual care services for PTSD through the VHA for 12 weeks after which time they will be offered the physical activity program for 12 weeks. 18 patients were randomized, of which 17 completed the study (included in analyses).
Arm/Group | Exercise | Usual Care Wait-List
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/17
Other Adverse Events (participants affected / at risk) | 0/31 | 0/17

LIMITATIONS AND CAVEATS:
The recruitment period started November 2015 and was originally planned to last 18 months, but was extended to 2 years due to various life events of the PI that caused delays in recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT02295995/Prot_SAP_000.pdf